CLINICAL TRIAL: NCT06441448
Title: potentiALS - A Multi-method Participatory Aproach to Identify Potentials in Improving Quality of Life Among Patients With Amyotrophic Lateral Sclerosis
Brief Title: potentiALS - Quality of Life Among Patients With Amyotrophic Lateral Sclerosis
Acronym: potentiALS
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Leipzig University Medical Center (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Professor, University of Leipzig
Other Study IDs: 01KG2321
Record Dates: First submitted 2024-01-05; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: participatory aproach; quality of life; psychotherapeutic program
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: case focus groups — The study is in a monocentric, exploratory, participatory study conceptualization phase. Within the study, a mixed-methods assessment involves various interview and group exercise formats among scientists, medical personnel, affected individuals, and their caregivers to develop components for a future psychotherapeutic program for ALS patients and their caregivers. Therapists provide an overview of therapy forms by presenting components based on format, content, and applied techniques. Case studies and focus groups are used for practical experience for the participants. Participants qualitatively assess the significance of therapeutic approaches and make a quantitative prioritization to establish a ranking of therapy components.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a rapidly progressing and disabling disease with the majority of patients dying 3-5 years after symptom onset. Given the high symptom burden, many patients and its caregivers are highly distressed. However, few programs to improve mental health for this patient group exist, and the sparse research implies that programs effective in other medical conditions may not be feasible in ALS patients. Therefore, it is highly needed to involve ALS patients, caregivers and medical staff as contributors into the development of such programs to meet the needs they really have.

The envisaged project has two aims: First, the investigators want to examine whether and how it is possible to involve ALS patients in the whole research process despite rapid disease progress and severe functional impairments. Second, the investigators are interested in how contributors (i.e., patients, caregivers and medical staff) would compile a concrete psychotherapeutic program, i.e., how they set priorities in terms of format, content and treatment techniques of such a program.

The investigators will closely collaborate with contributors across the whole project in designing the research process, planning assessment as well as interpreting and disseminating the findings. At the end of the study, the investigators will gather contributor feedback on their experience with the participatory approach.

Results will provide important information on how ALS patients can be effectively involved in psychosocial intervention research. Identified priorites regarding psychotherapeutic programs will serve as concrete starting points to develop and test a disease-specific program within a subsequent study.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurogenerative multi-systemic disease with various symptoms including weakness, cramps, pain, inappropriate affect or speech problems. ALS is inevitably fatal, with the majority of patients dying within 3-5 years after symptom onset as a result of ventilatory failure.

Given the symptom burden and the fatal nature of the disease, many patients are highly distressed. ALS patients show elevated rates of depressive symptoms and impaired quality of life, and levels of anxiety increase with progressing disease. About one third of patients suffer from moderate or severe hopelessness which in turn is associated with desire for hastened death.

The mental burden warrants effective psychological treatments to improve quality of life (QoL) among this patient group. However, few psychosocial interventions studies exist whose results do not allow for strong recommendations due to issues regarding methodology and acceptability. Recently, our own working group failed to apply a psychotherapy effective in palliative cancer patients to ALS patients (publication in preparation, see https://clinicaltrials.gov/ct2/show/NCT03975608).

Therefore, concepts feasible in other populations may not meet the specific needs of ALS patients. Indeed, various disease-specific facilitators have been identified such as flexible format, diseasespecific content tailoring, fostering of patient autonomy, but also barriers such as high effort in reaching and undergoing the intervention and functional decline. Based on such findings, psychotherapeutic programs for ALS patients should be co-designed within a participatory approach to overcome problems with feasibility and acceptability. However, the investigators identified only one study applying a similar approach; however, it was placed in a complete different health care context.

The investigators herein envisage a conceptual phase closely collaborating with various contributors, i.e., patients, caregivers and medical staff. The first objective is to assess the ability and benefit in collaborating with ALS patients in psychosocial intervention research. As second objective, contributors will prioritize their needs in psychological interventions regarding format, content and techniques. Results will be used in an exploratory trial to co-design a psychotherapeutic program ensuring good feasibility and acceptability.

The research questions of the first objective are the following:

1. How high is the response rate of contributors to be involved in this participatory project?
2. Which participative methods are applicable among ALS patients or need to be adapted?
3. How do contributors evaluate the possbility to collaborate in psychosocial intervention research?
4. What are the lessons learned and how can they be transferred to participatory psychosocial intervention research among severe (neurodegenerative) diseases?

   The main research questions related to the second objective are the following:
5. How do contributors prioritize treatment-related factors in format, content and techniques?
6. Which factor-specific barriers for feasibility and acceptability are anticipated by contributors?
7. What are the main findings to serve as starting point for co-designing a disease-specific treatment program within an exploratory future trial?

ELIGIBILITY:
Inclusion Criteria:

* patients met criteria for definite/laboratory-supported probable/clinically probable/possible familial or sporadic ALS (diagnostically synonymous with MND) or MND variants (progressive muscular atrophy or primary lateral sclerosis according to the revised El Escorial criteria
* ≥ 18 years old
* fluent in German
* ability to communicate thoughts and feelings
* ability to provide written consent
* anticipated remaining lifespan of ≥ 9 months.

Exclusion Criteria:

* under 18 years old
* had a clinical need for gastrostomy feeding or non-invasive ventilation
* had a diagnosis of dementia
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes 20 dyads of individuals affected by ALS and their caregivers, 4 expert patients, and 10 healthcare professionals.
  The recruitment is conducted through patient networks and personal contacts established by the patient representative and the project leader (e.g., within neuropalliative networks). The project leader will also invite medical personnel through his networks and in the course of his clinical work (e.g., within the "Clinic for Motor Neuron Diseases" at Leipzig University Hospital) to participate in the study. Affected individuals may also be invited to participate in the study by the project leader during their medical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | through study completion, an average of 1 year
  The investigators will assess the amount of eligible patients which are willing to participate in the study relative to the amount of patients who were invited to participate.

SECONDARY OUTCOMES:
Level of Quality of Life | through study completion, an average of 1 year
  Assessed by a questionnaire, the Amyotrophic Lateral Sclerosis Assessment Questionnaires - short form (ALSAQ-5). The total score across the 5 items, rated on a 4-point Likert scale, will be presented (range: 0 - 20). Higher values indicate higher quality of life.enable ranking of preferences as well as qualitative focus groups/interviews for in-depth analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Metelmann, PhD, Principal Investigator — Universitätsklinikum Leipzig
Locations (1):
- University Medical Center Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heyne S, Kuzmanova A, Esser P, Linse K, Gunther R, Mehnert-Theuerkauf A, Metelmann M. How can we reduce psychological burden for patients of amyotrophic lateral sclerosis and their family caregivers? - Insights from the participatory multi-method study "potentiALS". BMC Neurol. 2025 Oct 7;25(1):414. doi: 10.1186/s12883-025-04440-w. PMID 41057832